CLINICAL TRIAL: NCT06055231
Title: A Randomized Within-Subject Cross-Over Study to Compare Short-Term PK/PD Effects of Vaping THC-containing Liquids vs. Smoked Cannabis
Brief Title: PK/PD of Vaping THC-containing Liquids vs. Smoked Cannabis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: I 3409223; R01DA057228 (NIH)
Record Dates: First submitted 2023-09-07; First posted 2023-09-26 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1 (Vape followed by Joint) (Experimental): Patients receive a vape device with THC containing liquid and consume the provided amount in up to 10 minutes. 7 to 14 days later patients receive a cannabis joint and smoke the provided joint in up to 10 minutes. Patients also undergo blood sample collection throughout the study.
  Interventions: Behavioral: Vape device; Drug: Marijuana via joint
- Arm II (Joint followed by Vape) (Experimental): Patients receive a cannabis joint and smoke the provided joint in up to 10 minutes. 7 to 14 days later patients receive a vape device with THC containing liquid and consume the provided amount in up to 10 minutes. Patients also undergo blood sample collection throughout the study.
  Interventions: Behavioral: Joint; Drug: Marijuana via vape device

INTERVENTIONS:
Behavioral: Vape device — Consume THC via vape defice
  Other Names: Behavioral Conditioning therapy; Behavioral Modification
  Arms: Arm 1 (Vape followed by Joint)
Behavioral: Joint — Consume THC via joint
  Other Names: Behavior Conditioning Therapy; Behavior Modification
  Arms: Arm II (Joint followed by Vape)
Drug: Marijuana via vape device — Given via vape device
  Other Names: Cannibis
  Arms: Arm II (Joint followed by Vape)
Drug: Marijuana via joint — Given via joint
  Other Names: Cannibis
  Arms: Arm 1 (Vape followed by Joint)

SUMMARY:
We will conduct a randomized, within-subjects clinical study to compare short-term pharmacokinetic (PK) and pharmacodynamic (PD) effects of Δ9-tetrahydrocannabinol (THC) vaping liquids vs. smoked cannabis containing 6 equivalent standard THC units (5 mg THC=1 Standard THC Unit (STU)) in healthy community members who are current users of both products. While smoking cannabis remains the most common mode of THC use among adults and youth, alternative modes of delivery, such as Electronic Vaping Products (EVPs), are becoming increasingly popular for the delivery of cannabinoids. Declining cannabis risk perceptions, increasing normalization of cannabis, greater legal access and availability to cannabis, ease of administration, and ability to conceal vaped THC use have likely contributed to increasing prevalence of use throughout the population across all age groups. Comparing vaping THC containing liquids with smoking cannabis can serve as an important benchmark for evaluating the delivery and effects of THC vaping products and, their relative safety

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare the PK/PD profiles of delta-9 tetrahydrocannabinol (THC) from equivalent standard THC doses (30mg) administered as vaped THC liquid vs. smoked cannabis using a within-subject design.

SECONDARY OBJECTIVES:

I. Safety

PRIMARY OBJECTIVE:

I. Compare the PK/PD profiles of delta-9 tetrahydrocannabinol (THC) from equivalent standard THC doses (30mg) administered as vaped THC liquid vs. smoked cannabis using a within-subject design.

SECONDARY OBJECTIVES:

I. Safety

ELIGIBILITY:
Inclusion Criteria:

* Age >= 21 years of age
* Report concurrent use of commercial (medical or recreational) smoked cannabis and THC vaping cartridges for at least 3 months prior to enrollment
* Report smoking cannabis and THC- vaping liquid use at the potency level of the study product at least weekly (4x/month)
* Report of not currently trying to become pregnant (females). Women of childbearing potential must be willing to provide a urine sample and test negative prior to receiving any study-related products/procedures
* Willing to complete a THC saliva test to check for recent use (NarcoCheck Ref#:NCE-STHC-1) and semi -quantitative urinary tetrahydrocannabinol-carboxylic acid (THCA) rapid test (NarcoCheck® THC PreDosage) during baseline testing, prior to receiving any study-related products
* Participant must understand the investigational nature of this study and sign an Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* • Illegal or non-prescription drug use within the past 90 days. As detected by NacroCheck® Évolutive® (detection in human urine of the 12 most currently abused drugs) at the first session and prior to receiving any study product

  * Report 2 or more drinking occasions/week with 4 or more drinks/occasion
  * Report of daily nicotine use
  * Current or prior diagnosis of any psychotic disorders
  * Current or prior diagnosis of chronic heart conditions
  * Current or prior diagnosis of any respiratory condition
  * Pregnant or currently trying to become pregnant (females)
  * Detection level 4-5 (>300 ng/mL) from a semi-quantitative urinary THCA rapid test (NarcoCheck® THC PreDosage)
  * Unwilling or unable to follow protocol requirements
  * Any condition which in the Investigator's opinion deems the participant an unsuitable candidate for participation

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | From baseline to 360 minutes after consuming product
  Blood samples will be collected for plasma levels of THC. All individual pharmacokinetic (PK) parameters will be derived from plasma THC concentrations-versus-time data by non-compartmental analysis using Phoenix WinNonlin, corrected for baseline THC concentrations. Mean differences for each measure will be compared between the experimental (THC vaping) and active control (smoked cannabis) conditions, and by sex
Area under the plasma concentration time curve from 0-360 minutes ((AUC^0-360) | From baseline to 360 minutes after consuming product
  Blood samples will be collected for plasma levels of THC. All individual pharmacokinetic (PK) parameters will be derived from plasma THC concentrations-versus-time data by non-compartmental analysis using Phoenix WinNonlin, corrected for baseline THC concentrations. Mean differences for each measure will be compared between the experimental (THC vaping) and active control (smoked cannabis) conditions, and by sex.
Time to maximum concentration of THC in plasma (Tmax) | From baseline to 360 minutes after consuming product
  Blood samples will be collected for plasma levels of THC.All individual pharmacokinetic (PK) parameters will be derived from plasma THC concentrations-versus-time data by non-compartmental analysis using Phoenix WinNonlin, corrected for baseline THC concentrations. Mean differences for each measure will be compared between the experimental (THC vaping) and active control (smoked cannabis) conditions, and by sex.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 360 minutes after consuming product
  Number of subjects who experienced an adverse event during the study .
Puffing behaviors | Through study completion, an average of 14 days
  Measure changes in subject puffing behavior by mean number of puffs and duration
Short term effects of THC | Through Study completion, an average of 14 days
  The Drug Effect Questionnaire (DEQ) rates sixteen component items using a visual analog scale (0-100) to examine drug effects pre- and post-use.
Cognitive Performance as assessed by the Digit Symbol Substitution Task (DSST) | Through study completion, an average of 14 days
  computerized sensitive and valid assessment of cognitive dysfunction that correlates with real-world functional ability to complete daily tasks. The outcome is the total number of correct responses.
Paced Auditory Serial Addition Task (PASET) | Through study completion , an average of 14 days
  a validated measure used to assess attention, concentration, working memory, and information processing.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Smith, Principal Investigator — Roswell Park Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: Undecided